CLINICAL TRIAL: NCT04513327
Title: New Model of Short-term Rehabilitation Exercise Training Using Digital Healthcare System in Patients With Anterior Cruciate Ligament Reconstruction; Randomized Controlled Study
Brief Title: Rehabilitation Exercise Using Digital Healthcare System in Patients With Anterior Cruciate Ligament Reconstruction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Collaborators: Ministry of Health, Republic of Korea (Other Government)
Responsible Party: Principal Investigator, Jae-Young Lim, Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B-2005/612-001(3)
Record Dates: First submitted 2020-08-09; First posted 2020-08-14 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2022-01

CONDITIONS: Anterior Cruciate Ligament Injuries
Keywords: Anterior Cruciate Ligament Reconstruction; Post-Operative Rehabilitation; Digital Healthcare System
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital Healthcare System Rehabilitation (Experimental)
  Interventions: Device: Rehabilitation using Digital Healthcare System (Uincare Homeplus)
- Conventional Rehabilitation (Active Comparator)
  Interventions: Other: Conventional Rehabilitation

INTERVENTIONS:
Device: Rehabilitation using Digital Healthcare System (Uincare Homeplus) — Uincare Homeplus is a device using infrared, kinect camera and motion capture technology to track 3D motion of the patients' posture and joint articulations. It also has embedded exercise training software dedicated to anterior cruciate ligament reconstruction post-op rehabilitation at home.
  Home-based self-rehabilitation using brochure for 2 weeks post surgery (same as the active comparator)
  Home-based self-rehabilitation using digital healthcare system(Uincare Homeplus) for 2 to 12 weeks post surgery.
  Other Names: Uincare Homeplus
  Arms: Digital Healthcare System Rehabilitation
Other: Conventional Rehabilitation — Home-based self-rehabilitation using brochure for 12 weeks post surgery.
  Arms: Conventional Rehabilitation

SUMMARY:
The study aims to examine the effect of short-term rehabilitation exercise support using digital healthcare system (Uincare homeplus) in the patients with anterior cruciate ligament reconstruction. The study is a two-arm prospective randomized controlled study comparing the effect of rehabilitation exercise digital healthcare system at home with conventional brochure-based home exercise. Limb Symmetry Index (LSI), Pain (using Numerical rating scale), knee joint range of motion (ROM), lower extremities motor power (using Manual muscle test), International Knee Documentation Committee (IKDC) and quality of life using EQ-5D-5L will be evaluation on enrollment, 2-weeks, 6-weeks, 12-weeks and 24-weeks after enrollment.

DETAILED DESCRIPTION:
Anterior cruciate ligament(ACL) is a vital structure in the knee maintaining the stability and due to increased population engaging in sports activities, the ACL injury is becoming more prevalent among young adults. Rehabilitation after ACL reconstruction is essential to restore knee function and many factors including age, degree of sports activities engagement, weight bearing should be considered when organizing rehabilitation programs. Knee joint stiffness and weakness of knee flexor/extensor muscles are common problems following the surgery which are related to improper rehabilitation after ACL reconstructions.

Current method of post-operative rehabilitation is home-based self rehabilitation using brochure, combined with one or two times of education at the hospital before discharge. Patients often find difficulty in doing rehabilitation by themselves at home without supervision which resulted in decreased compliance.

With development of technologies using multi-motion sensor and AR(augmented-reality) system, the investigators have developed a digital healthcare system(Uincare Homeplus) which can supplement patients' rehabilitation at home by giving them proper instructions as well as feedback. In this prospective randomized controlled study, the investigators aim to compare the efficacy of the newlydeveloped digital healthcare system with conventional rehabilitation program.

ELIGIBILITY:
Inclusion Criteria:

* Patient who had anterior cruciate ligament reconstruction surgery
* Patient who is discharged to home after surgery

Exclusion Criteria:

* Patient who had previous history of anterior cruciate ligament reconstruction surgery in the past 6 months.
* Patient who had undergone bilateral anterior cruciate ligament reconstruction surgery.
* Patient who has knee joint disorders (rheumatoid arthritis, osteoarthritis) other than anterior cruciate ligament injury.
* Patient who has neurological deficit or infection in the affected knee joint.
* Patient who has severe comorbidity that inhibits exercise.
* Patient who cannot participate in post surgery rehabilitation

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-07-30 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline Limb Symmetry Index (LSI) of lower extremities | Enrollment, 2-weeks, 6-weeks, 12-weeks, 24-weeks
  LSI(%) = (involved limb knee flexor and extensor manual muscle test score / uninvolved limb knee flexor and extensor manual muscle test score * 100). LSI ranges from 0-100 with higher score meaning better limb symmetry.

SECONDARY OUTCOMES:
Numerical Rating Scale (NRS) on the affected knee | Enrollment, 2-weeks, 6-weeks, 12-weeks, 24-weeks
  Evaluation of pain of the affected shoulder using numerical rating scale (0-10, with score 0 indicating no pain). Higher score meaning worse pain.
Range of Motion (ROM) on the affected knee | Enrollment, 2-weeks, 6-weeks, 12-weeks, 24-weeks
  Evaluation of change of ROM in the affected knee from baseline to 24 weeks
Manual Muscle Test (MMT) on the affected lower extremities | Enrollment, 2-weeks, 6-weeks, 12-weeks, 24-weeks
  Evaluation of change of MMT in the affected lower extremities from baseline to 24 weeks. Affected lower extremity MMT ranges from 0-25 with higher score meaning better motor power.
International Knee Documentation Committee (IKDC) score on the affected knee | Enrollment, 2-weeks, 6-weeks, 12-weeks, 24-weeks
  IKDC score is a self-reported measure, 18 items (7 on symptoms, 1 on participation in sports, 9 on daily activities, and 1 on current knee function). IKDC score ranges from 0-100, with higher score meaning better function.
Quality of Life using EQ-5D-5L | Enrollment, 2-weeks, 6-weeks, 12-weeks, 24-weeks
  Evaluation of quality of life using EQ-5D-5L. This scale is numbered from -0.066 to 0.904. Lower value means worse quality of life.

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Samsung Medical Center, Seoul, Gangnam-gu
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lim JY, Yu HJ, Kim SH, Lee JI, Lim JY, Wang JH, Hwang JH. Effectiveness of In-Home, Augmented Reality-Based Telerehabilitation After Anterior Cruciate Ligament Reconstruction: A Randomized Controlled Trial. Orthop J Sports Med. 2024 Oct 15;12(10):23259671241271729. doi: 10.1177/23259671241271729. eCollection 2024 Oct. PMID 39415796